CLINICAL TRIAL: NCT05894512
Title: Analysis of T- and B-Cell Subpopulations in Patients With Primary Membranous Nephropathy
Brief Title: Analysis of T- and B-Cell Subpopulations in Membranous Nephropathy
Status: Active, not recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Mirioglu, Principal Investigator, Istanbul University
Other Study IDs: 2023/887
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Membranous Nephropathy; Membranous Nephropathy - PLA2R Induced; Membranous Nephropathy - THSD7A Induced
Keywords: membranous nephropathy; rituximab; flow cytometry; immunophenotyping; PLA2R
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood samples from the volunteers will be taken into 20 ml EDTA, heparinized and dry tubes. Blood samples taken into a 10 ml dry tube will be centrifuged at 3000 rpm for 10 minutes. After the process, the separated serum will be placed in Eppendorf tubes (microcentrifuge tubes) and frozen at -20°C for 48 hours, and then transferred to deep freezers to be stored at -80°C.
  Peripheral blood mononuclear cells (PBMCs) will be obtained from blood samples by Ficoll concentration gradient centrifugation method. PBMCs collected after centrifugation will be suspended with fetal bovine serum (FBS). Cells in FBS medium will be taken into cryotubes, frozen in liquid nitrogen (-196°C) by adding dimethyl sulfoxide and stored until the laboratory studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study Group (Primary Membranous Nephropathy): Patients with biopsy-proven primary membranous nephropathy will be included (n=18).
  Samples will be collected from patients diagnosed with primary MN before starting conventional immunosuppressive therapy with calcineurin inhibitors (CNI) and corticosteroids (CS) and at 3, 6, 12, 18 and 24 months after starting the treatment.
  In case of failure after treatment with CNIs and CS treatment, rituximab (RTX) is used. If patient switches to RTX, samples will be taken before and 1, 3, 6, 12, 18, and 24 months after the first dose of RTX.
  If relapse occurs, sampling will be done regardless of the timing.
  Treatment decisions will solely be made in line with the guidelines, and there will be no intervention.
- Control Group 1 (IgA Nephropathy): After the patient group sampling is completed, a diseased control group will be formed from patients with primary IgA nephropathy according to the distribution of age and sex (n=15).
  Samples will be collected from the patients for one time only (cross-sectional sampling).
- Control Group 2 (Healthy Volunteers): After the patient group sampling is completed, a healthy control group will be formed from healthy volunteers according to the distribution of age and sex (n=15).
  Samples will be collected from healthy volunteers for one time only (cross-sectional sampling).

SUMMARY:
The aim of this observational study is to provide analysis of T and B lymphocyte subgroups in peripheral blood samples of patients with primary membranous nephropathy (MN). A search for disease-related circulating antibodies [anti-phospholipase A2 receptor antibody (anti-PLA2R) and anti-thrombospondin type 1 domain-containing 7A antibody (anti-THSD7A)] in patients' sera is also planned.

The main questions to answer are:

1. What is the relationship of these cell populations and their distribution during follow-up with treatment, treatment responses, and relapses?
2. What is the relationship of the cell populations with anti-PLA2R (or anti-THSD7A) antibody levels?

Participants will provide peripheral venous blood samples at pre-designated regular intervals.

The research team will compare results of the primary MN group with two control groups (IgA nephropathy and healthy volunteer groups) to see if the findings are specific for primary MN.

DETAILED DESCRIPTION:
Primary membranous nephropathy (MN), which is one of the most common causes of nephrotic syndrome in adults, is an autoimmune disease characterized with remissions and exacerbations. About half of the patients who do not go into remission progress to end-stage kidney disease.

In recent years, a lot of progress has been made in the fields of nephrology and immunology regarding primary MN. The process, which began with the detection of autoantibodies against the M-type phospholipase A2 receptor (PLA2R) in approximately 70% of the patients, continued with the discovery of new molecules for diagnosis and follow-up. However, despite all these advances, studies based on the analysis of peripheral blood mononuclear cells in patients with primary MN are very few: Rosenzwajg et al. analyzed lymphocyte subgroups in 25 MN patients and 27 healthy controls, and showed that regulatory T cells were significantly decreased in patients, naive B cells were increased, and memory B cells were decreased (Rosenzwajg et al. Kidney Int 2017). In 2020, Cantarelli et al. performed an extensive analysis in 30 patients with MN, showing that regulator B cells were increased in the MN group (Cantarelli et al. Kidney Int Rep 2020). These studies were generally cross-sectional or sampling was performed at a maximum of 6 months of follow-up. More studies based on long-term follow-up are needed.

Therefore, the aim of this observational study is to provide analysis of T and B lymphocyte subgroups in peripheral blood samples of patients with primary MN. A search for disease-related circulating antibodies [anti-phospholipase A2 receptor antibody (anti-PLA2R) and anti-thrombospondin type 1 domain-containing 7A antibody (anti-THSD7A)] in patients' sera is also planned. It is designed to investigate the relationship of these cell populations and their distribution during follow-up with treatment, treatment responses, and relapses. The relationship of cell populations with antibody levels over time will also be examined.

By investigating the distribution of T and B lymphocyte subgroups in patients with primary MN during the follow-up, and its relationship with treatment, treatment responses, and relapses, it is expected to better elucidate the pathogenesis of the disease and to detect cell changes suggestive of remission and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of primary membranous nephropathy (patient group).
* Having a diagnosis of primary IgA nephropathy (diseased control group).
* Being healthy (healthy control group).
* Agreeing to participate in the research (informed consent).

Exclusion Criteria:

* Refusing to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven membranous nephropathy (study group) and IgA nephropathy (control group).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of T- and B-cell subpopulations | 2 years
  Distribution of T- and B-cell subpopulations will be evaluated with flow cytometry throughout the 2-year follow-up process.

SECONDARY OUTCOMES:
Complete remission | 2 years
  Reduction of proteinuria to <0.3 g/g or g/day, stable serum creatinine, and serum albumin >3.5 g/dl.
Partial remission | 2 years
  Reduction of proteinuria to 0.3-3.5 g/g or g/day with an at least a 50% decrease from the baseline.
Relapse | 2 years
  Proteinuria of at least 3.5 g/g or g/day after complete or partial remission has been reached.
Composite kidney outcome | 2 years
  Initiation of kidney replacement therapies (hemodialysis, peritoneal dialysis or kidney transplantation), development of stage 5 chronic kidney disease (eGFR <15 ml/min/1.73 m2), or at least a 50% loss in eGFR.

OTHER OUTCOMES:
Serum anti-PLA2R IgG antibody levels | 2 years
  Serum anti-PLA2R IgG antibody levels will be evaluated with enzyme-linked immunosorbent assay (ELISA) throughout the 2-year follow-up process.
Serum anti-THSD7A IgG antibody levels | 2 years
  In PLA2R-negative patients, serum anti-THSD7A IgG antibody levels will be evaluated with indirect immunofluorescence test (IIFT) throughout the 2-year follow-up process.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Adin Cinar, PhD, Study Chair — Istanbul University; Safak Mirioglu, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenzwajg M, Languille E, Debiec H, Hygino J, Dahan K, Simon T, Klatzmann D, Ronco P. B- and T-cell subpopulations in patients with severe idiopathic membranous nephropathy may predict an early response to rituximab. Kidney Int. 2017 Jul;92(1):227-237. doi: 10.1016/j.kint.2017.01.012. Epub 2017 Mar 15. PMID 28318628
- [Background] Cantarelli C, Jarque M, Angeletti A, Manrique J, Hartzell S, O'Donnell T, Merritt E, Laserson U, Perin L, Donadei C, Anderson L, Fischman C, Chan E, Draibe J, Fulladosa X, Torras J, Riella LV, La Manna G, Fiaccadori E, Maggiore U, Bestard O, Cravedi P. A Comprehensive Phenotypic and Functional Immune Analysis Unravels Circulating Anti-Phospholipase A2 Receptor Antibody Secreting Cells in Membranous Nephropathy Patients. Kidney Int Rep. 2020 Aug 1;5(10):1764-1776. doi: 10.1016/j.ekir.2020.07.028. eCollection 2020 Oct. PMID 33102969